CLINICAL TRIAL: NCT05239715
Title: Evaluation of Three SS-OCT and One PCI Optical Biometers in Eyes With Dense Cataract: Benefit of Use of the Enhance Retina Visualization Mode
Brief Title: Evaluation of Three SS-OCT and One PCI Optical Biometers in Eyes With Dense Cataract
Acronym: BIO-CAT-DENSA
Status: Completed | Type: Observational
Sponsor: OFTALVIST (Oftalmología Vistahermosa S.L) (Industry)
Collaborators: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: BIO-CAT-DENSA
Record Dates: First submitted 2022-02-03; First posted 2022-02-15 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Optical Biometer, Cataracts
Keywords: optical biometer, cataracts
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Ocular biometry — Biometry using swept-source OCT Argos, swept-source OCT IOLMaster 700, swept-source OCT Anterion, PCI Pentacam AXL, OcuScan RxP and Itrace measurement

SUMMARY:
To describe and compare the acquisition rate between different biometers in eyes with advanced cataracts

DETAILED DESCRIPTION:
To describe and compare the acquisition rate between different biometers in eyes with advanced cataracts

ELIGIBILITY:
Inclusion Criteria:

* LOCS III cataract classification with a grade of ≥3 for nuclear, cortical or posterior subcapsular.
* DLI index, from the ITrace device, should be ≤ 5.

Exclusion Criteria:

* Previous continuous contact lens wear
* Ocular trauma
* Intraocular lens surgery
* Poor fixation
* Corneal disease (i.e. keratoconus)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with dense cataracts.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
To describe and compare the acquisition rate between different biometers in eyes To describe and compare the acquisition success rate between different biometers in eyes with advanced cataracts | 6 months
  Acquision succes rate is indicated by a percentage, from 0% to 100%. The biometer can obtain (success) or not (failure) the measurement. This value will be indicated for each biometer.

SECONDARY OUTCOMES:
To describe the correlation of success rate and Dysfunctional Lens Index (DLI, iTrace) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Tañá, Dr., Principal Investigator — Oftalmología Vistahermosa SL
Locations (1):
- Oftalmología Vistahermosa SL, Alicante, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tana-Rivero P, Aguilar-Corcoles S, Tana-Sanz P, Tana-Sanz S, Montes-Mico R. Axial length acquisition success rates and agreement of four optical biometers and one ultrasound biometer in eyes with dense cataracts. Eye Vis (Lond). 2023 Sep 1;10(1):35. doi: 10.1186/s40662-023-00352-3. PMID 37653460